CLINICAL TRIAL: NCT00363610
Title: A Multicenter, Open-Label, Phase I Study Evaluating the Safety and Tolerability of Intravenous Pegaspargase in Combination With Intravenous Gemcitabine HCl in the Treatment of Advanced and/or Metastatic Solid Tumors and Lymphoma
Brief Title: A Study Evaluating IV Oncaspar® and IV Gemzar® in the Treatment of Solid Tumors and Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: No recommended Phase II dose was determined.
Sponsor: Enzon Pharmaceuticals, Inc. (Industry)
Responsible Party: Enzon Pharmaceuticals, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EZ-002-001
Record Dates: First submitted 2006-08-09; First posted 2006-08-15 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Tumors; Lymphoma
Keywords: Advanced and/or Metastatic Solid Tumors and Lymphoma
MeSH Terms: conditions — Neoplasms; Lymphoma | interventions — pegaspargase; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Oncaspar & Gemzar; advanced and/or solid tumors and lymphoma

SUMMARY:
This study will research the side effects of pegaspargase (pronounced "peg-as-par-gase"); its brand name is ONCASPAR® when it is used with another FDA-approved cancer treatment (chemotherapy) drug called gemcitabine HCl (pronounced "gem-site-a-bean"; its brand name is GEMZAR®.

DETAILED DESCRIPTION:
The purpose of this research study is for the study's sponsor, Enzon Pharmaceuticals, Inc. ("Enzon"), to learn more about its drug pegaspargase. Pegaspargase is the drug's scientific or generic name. Because it is already approved by the Food and Drug Administration (FDA), it also has a brand name - ONCASPAR®. It is approved by the FDA for the treatment of a type of leukemia (cancer of white blood cells). However, pegaspargase is not approved by the FDA for treatment of the cancer in this study. This study will research the side effects of pegaspargase when it is used with another FDA-approved cancer treatment (chemotherapy) drug called gemcitabine HCl; its brand name is GEMZAR®. It is approved for the treatment of patients with cancer of the pancreas and of patients with breast cancer. However, gemcitabine is not approved by the FDA for treatment of any other types of cancer.

In addition, the combination of pegaspargase and gemcitabine for solid tumors and lymphoma in this study is investigational. This type of study treatment is called a "combination treatment" or a "combination study." The information (research data) from this study will be used by Enzon to plan other "combination" research studies with pegaspargase plus gemcitabine for the treatment of certain cancers.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding the protocol requirements and risks and providing written informed consent.
* Histologically or cytologically confirmed diagnosis of advanced and/or metastatic solid tumor or lymphoma (Hodgkin's or non-Hodgkin's), and have either failed primary treatment or there is no available standard treatment.
* Prior standard therapy was not effective, or no known therapy will extend survival or provide benefit.
* Measurable or evaluable disease.
* Age 18 years or older.
* Score of 0-2 on the Eastern Cooperative Oncology Group (ECOG) performance scale.
* Absolute neutrophil count (ANC)≥ 1500/μL.
* Platelet count ≥ 100,000/μL.
* Hemoglobin ≥ 9.0 g/dL.
* Fibrinogen ≥ 0.75x the lower limit of normal (LLN), and PT, PTT, and INR ≤ 1.5x the upper limit of normal (ULN).
* Serum creatinine ≤ 1.5 mg/dL or creatinine clearance ≥ 60 mL/min.
* Total bilirubin ≤ 1.5 mg/dL.
* Transaminases (AST, ALT) ≤ 2.5x the upper limit of normal (ULN) (may be ≤ 5.0x ULN if due to metastatic disease in the liver).
* Amylase and lipase levels are within normal limits.

Any subject who has given informed consent to participate in the clinical study and who meets all entry criteria for the study may participate in the tumor analysis part of the study.

Exclusion Criteria:

* Subjects meeting any of the following exclusion criteria will not be eligible for enrollment.
* Concurrent serious medical illness that could potentially interfere with protocol compliance.
* Has pancreatitis or a history of pancreatitis, not related to pancreatic cancer.
* Has a coagulopathy or a history of coagulopathy.
* Known chronic infectious disease, such as AIDS or hepatitis (screening for hepatitis and HIV will not be performed).
* Positive screening pregnancy test or is breast-feeding.
* Female or male subject of reproductive capacity unwilling to use methods appropriate to prevent pregnancy during the course of this protocol.
* Known or clinically suspected active brain metastases.
* Received pegaspargase (Oncaspar®, PEG-L-asparaginase) or any asparaginase or asparaginase-containing drug, at any time prior to this study.
* Received prior chemotherapy, immunotherapy or an investigational agent regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-07; Primary Completion 2007-11 (Actual); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
The primary objectives of this Phase 1 study of pegaspargase in combination with gemcitabine are to determine the maximum tolerated dose of IV pegaspargase when administered with gemcitabine
and to determine the recommended Phase 2 dose of pegaspargase

SECONDARY OUTCOMES:
The secondary objectives of this study are to evaluate the safety and tolerability of the combination study treatment
to determine the PD/PK profile and immunogenicity of pegaspargase
to determine the PK profile of gemcitabine when administered in combination with pegaspargase
and to detect preliminary evidence of tumor

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - TGen Clinical Research Services at Scottsdale Healthcare, Scottsdale, Arizona
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cancer Therapy & Research Center, Institute for Drug Development, San Antonio, Texas